CLINICAL TRIAL: NCT00114491
Title: Rosuvastatin Affecting Aortic Valve Endothelium - RAAVE
Brief Title: Rosuvastatin Affecting Aortic Valve Endothelium
Status: Completed | Type: Observational
Sponsor: Hospital Pedro Hispano (Other)
Collaborators: Northwestern University (Other)
Other Study IDs: 22352
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Last update posted 2006-10-31 (Estimated); Status verified 2006-10

CONDITIONS: Atherosclerosis; Hypercholesterolemia
Keywords: Aortic Stenosis; Statins; Hypercholesterolemia
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Aortic Valve Stenosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: Rosuvastatin

SUMMARY:
Recent studies support the hypothesis that aortic stenosis (AS) develops due to atherosclerosis affecting the aortic valve endothelium. The study's aim was to assess Rosuvastatin on the hemodynamic progression and inflammatory markers of AS by treating low-density lipoprotein (LDL) in patients with AS according to the National Cholesterol Education Program Adult Treatment Panel III (NCEP-ATPIII) guidelines for one year.

DETAILED DESCRIPTION:
Background: Recent retrospective studies support the hypothesis that statins slow the progression of aortic stenosis. The aim of this study was to assess the effect of Rosuvastatin on hemodynamic progression of aortic stenosis by treating patients with aortic stenosis and elevated LDL-cholesterol for 18 months.

Methods: We performed an open-label, prospective study evaluating 121 consecutive patients with asymptomatic moderate to severe aortic stenosis (AVA≥ 1.0 cm2), (mean age 73.7±8.9 years; 57 men and 64 women), treated with and without Rosuvastatin according to the NCEP-ATPIII guidelines. Echocardiographic, serum lipid, and inflammatory markers were measured at baseline and every 6 months for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic AS
* Normal ejection fraction
* Elevated LDL >130 mg/dl

Exclusion Criteria:

* Echocardiographic evidence of rheumatic mitral valve disease,
* Previous statin therapy,
* Congenital heart disease (bicuspid aortic valve),
* Subaortic obstruction,
* Creatinine ≥ 2,0 mg/dl (to avoid the potential confounder of an elevated serum [CaP04]),
* Evidence of liver disease,
* Greater than mild aortic regurgitation and previous aortic valve surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-09; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Moura, Principal Investigator — Hospital Pedro Hispano
Locations (1):
- Hospital Pedro Hispano, Porto, Portugal

REFERENCES:
- [Result] Rajamannan NM, Subramaniam M, Stock SR, Stone NJ, Springett M, Ignatiev KI, McConnell JP, Singh RJ, Bonow RO, Spelsberg TC. Atorvastatin inhibits calcification and enhances nitric oxide synthase production in the hypercholesterolaemic aortic valve. Heart. 2005 Jun;91(6):806-10. doi: 10.1136/hrt.2003.029785. PMID 15894785
- [Result] Makkena B, Salti H, Subramaniam M, Thennapan S, Bonow RH, Caira F, Bonow RO, Spelsberg TC, Rajamannan NM. Atorvastatin decreases cellular proliferation and bone matrix expression in the hypercholesterolemic mitral valve. J Am Coll Cardiol. 2005 Feb 15;45(4):631-3. doi: 10.1016/j.jacc.2004.11.023. No abstract available. PMID 15708716
- [Result] Rajamannan NM. Is it time for medical therapy for aortic valve disease? Expert Rev Cardiovasc Ther. 2004 Nov;2(6):845-54. doi: 10.1586/14779072.2.6.845. PMID 15500430
- [Result] Rajamannan NM, Edwards WD, Spelsberg TC. Hypercholesterolemic aortic-valve disease. N Engl J Med. 2003 Aug 14;349(7):717-8. doi: 10.1056/NEJMc031360. No abstract available. PMID 12917318
- [Result] Otto CM. Why is aortic sclerosis associated with adverse clinical outcomes? J Am Coll Cardiol. 2004 Jan 21;43(2):176-8. doi: 10.1016/j.jacc.2003.10.027. No abstract available. PMID 14736433
- [Result] Rajamannan NM, Otto CM. Targeted therapy to prevent progression of calcific aortic stenosis. Circulation. 2004 Sep 7;110(10):1180-2. doi: 10.1161/01.CIR.0000140722.85490.EA. No abstract available. PMID 15353511
- [Result] Rajamannan NM, Subramaniam M, Rickard D, Stock SR, Donovan J, Springett M, Orszulak T, Fullerton DA, Tajik AJ, Bonow RO, Spelsberg T. Human aortic valve calcification is associated with an osteoblast phenotype. Circulation. 2003 May 6;107(17):2181-4. doi: 10.1161/01.CIR.0000070591.21548.69. Epub 2003 Apr 28. PMID 12719282
- [Derived] Moura LM, Ramos SF, Zamorano JL, Barros IM, Azevedo LF, Rocha-Goncalves F, Rajamannan NM. Rosuvastatin affecting aortic valve endothelium to slow the progression of aortic stenosis. J Am Coll Cardiol. 2007 Feb 6;49(5):554-61. doi: 10.1016/j.jacc.2006.07.072. Epub 2007 Jan 22. PMID 17276178